CLINICAL TRIAL: NCT02633982
Title: Registry Study on the Effectiveness of Rivaroxaban in Patients With Non-valvular Atrial Fibrillation Managed by General Practitioners(GENERAL Study)
Brief Title: GENERAL;GENeral Practitioners and Embolism pRevention in NVAF Patients Treated With RivAroxaban:reaL-life Evidence
Acronym: GENeRAL
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Japan Cardiovascular Research Foundation (Other)
Responsible Party: Sponsor
Other Study IDs: GENeRAL/J
Record Dates: First submitted 2015-12-09; First posted 2015-12-17 (Estimated); Last update posted 2015-12-17 (Estimated); Status verified 2015-11

CONDITIONS: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: Yes

SUMMARY:
In atrial fibrillation patients,anticoagulant therapy with warfarin has an excellent stroke preventive. Meantime,Warfarin may also increase the risk of hemorrhagic events. Considering this,warfarin is a drug which puts a great burden on patients and medical providers.

With the population aging, the number of non-valvular atrial fibrillation patients is increasing, and a necessity that not only specialist but also general practitioners. Anticoagulant therapy with warfarin is not easy for general practitioners and is not commonly used among general practioners. In such circumstances, Rivaroxaban,a new oral direct factor Xa inhibitor,has become available. Rivaroxaban is administrated once a day and exert an anti- coagulant effect soon after administration. It hardly reacts with foods or other drugs and therefore does not require regular monitoring. GENERAL study is to investigate the effectiveness of stroke and systemic embolism in non-valvular atrial fibrillation patients when it is prescribed by general practioners in real life settings.

ELIGIBILITY:
Inclusion Criteria:

* Non-valvular atrial fibrillation patient who are prescribed Rivaroxaban by General practitioners

Exclusion Criteria:

* Patients are contraindicated for rivaroxaban
* Patients judged as inappropriate for this study by investigators

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 5,000
Sampling Method: Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2015-09; Primary Completion 2018-10 (Estimated); Study Completion 2018-10 (Estimated)

PRIMARY OUTCOMES:
Composite of symptomatic stroke (ischemic/hemorrhagic) and systemic embolism | up to 1.5 years(max 3 years)

SECONDARY OUTCOMES:
Major bleeding events (adapted ISTH standard) | up to 1.5 years(max 3 years)
Non-major bleeding events(without Major Bleeding complications) | up to 1.5 years(max 3 years)
Composite of symptomatic stroke(ischemic or hemorrhagic),systemic embolism,myocardial infarction/unstable angina pectoris and cardiovascular death | up to 1.5 years(max 3 years)
Symptomatic stroke (ischemic or hemorrhagic) | up to 1.5 years(max 3 years)
Symptomatic ischemic stroke | up to 1.5 years(max 3 years)
Symptomatic hemorrhagic stroke | up to 1.5 years(max 3 years)
Systemic embolism | up to 1.5 years(max 3 years)
Acute myocardial infarction/unstable angina pectoris | up to 1.5 years(max 3 years)
Cardiovascular death | up to 1.5 years(max 3 years)
Deep vein thrombosis/pulmonary thromboembolism | up to 1.5 years(max 3 years)
Transient ischemic attack | up to 1.5 years(max 3 years)
Percutaneous coronary intervention /coronary artery bypass grafting | up to 1.5 years(max 3 years)
All cause death | up to 1.5 years(max 3 years)
Comparison of primary outcome (composite of symptomatic stroke(ischemic/hemorrhagic) and systemic embolism) rate and Major Bleeding complications (adapted ISTH standard)rate between EXPAND study and FUSHIMI AF registry | up to 1.5 years(max 3 years)
Adverse Event excluding hemorrhagic events | up to 1.5 years(max 3 years)
Patients adherence related with stroke or systemic embolism | up to 1.5 years(max 3 years)
Correlation with CHADS2 score or other risk factors and outcome events in Japanese patients who administered Rivaroxaban | up to 1.5 years(max 3 years)

CONTACTS AND LOCATIONS:
Locations (1):
- Japan Cardiovascular Research Foundation, Suita, Osaka, Japan

REFERENCES:
- [Derived] Matsui K, Kusano K, Akao M, Tsuji H, Hiramitsu S, Hatori Y, Odakura H, Ogawa H. Observational study of frailty in older Japanese patients with non-valvular atrial fibrillation receiving anticoagulation therapy. Sci Rep. 2024 Jun 22;14(1):14423. doi: 10.1038/s41598-024-65237-4. PMID 38909144